CLINICAL TRIAL: NCT00390598
Title: A Single Blind, Single Centre, Parallel Group, Randomized Controlled Trial Comparing PEG Solution (Laxabon®) 4L Versus Senna Glycoside (Pursennid® Ex-Lax) 36mg and PEG Solution (Laxabon®) 2L for Large Bowel Cleansing Prior to Colonoscopy
Brief Title: PEG Solution (Laxabon®) 4L Versus Senna Glycoside (Pursennid® Ex-Lax) 36mg and PEG Solution (Laxabon®) 2L for Large Bowel Cleansing Prior to Colonoscopy
Acronym: TARE-05-073M
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Markku Haapamäki, Umea University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TARE-05-073M
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2008-12

CONDITIONS: Colonoscopy
Keywords: colonoscopy; large bowel preparation; bowel cleansing; randomized controlled trial
MeSH Terms: interventions — Sennosides

ARMS (2):
- senna 36 mG + PEG 2L (Active Comparator): Bowel preparation with senna tablets 36 mG and PEG 2L prior to colonoscopy.
  Interventions: Drug: senna glycoside 36 mg and PEG (solution given 2 L)
- 4 L PEG (Active Comparator): Bowel preparation with 4 L PEG prior to colonoscopy.
  Interventions: Drug: PEG (solution given 4 L)

INTERVENTIONS:
Drug: PEG (solution given 4 L)
  Other Names: Laxabon (R) =PEG solution
  Arms: 4 L PEG
Drug: senna glycoside 36 mg and PEG (solution given 2 L)
  Other Names: Pursennid ExLax (R)= senna; Laxabon (R)= PEG solution
  Arms: senna 36 mG + PEG 2L

SUMMARY:
The trial compares Laxabon® 4L versus Pursennid® Ex-Lax 36mg and 2L Laxabon® for large bowel cleansing prior to colonoscopy allocating patients planned for colonoscopy to one of the two cleansing regimens.

DETAILED DESCRIPTION:
Effective large bowel cleansing prior to colonoscopy is still not achieved in all cases that undergo the procedure. The use of balanced electrolyte-polyethylene glycol (PEG) solution have improved the cleansing results and shortened the time needed for preparing the bowel. The problem with using PEG solution alone is the relatively large volume of the solution that the patients need to drink. The recommendation is to drink the solution until diarrhea fluid is clear and often 4 L or more is needed. Many patients refuse to drink the sufficient volume needed to get a clean colon. The large volume load can be a risk to patients suffering from renal and/or heart insufficiency.

Good results of bowel cleansing have also been reported with sodium phosphate solution or tablets. The fluid volume needed to drink along with sodium phosphate is generally no problem but this regimen causes electrolyte disturbances that usually are subclinical and of no significance but in patients with renal or heart insufficiency the sodium phosphate is contraindicated due to the risk of serious electrolyte disturbances.

Several combinations of stimulant laxatives with PEG solution have been tested before and the actual combination has been compared in one randomized study(1). Low-volume PEG plus sennosides preparation was better tolerated but it was not as effective as standard large-volume PEG.

PEG solution (Laxabon®) 4L is used for large bowel cleansing in many centers in Sweden and is the standard regimen used in our colonoscopy unit. In this study we compare this standard regimen with senna glycoside (Pursennid® Ex-Lax) 36mg (tablets) taken orally in the night before the colonoscopy and 2L Laxabon® solution orally starting to drink the solution four hours prior to the colonoscopy.

The result of large bowel cleansing is evaluated during the colonoscopy according to two separate validated scoring methods (Aronchick and Ottawa scores). Abdominal symptoms, discomfort, subjective grading of how hard/easy it was to complete the cleansing program and extra costs are evaluated with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo elective complete colonoscopy as an outpatient
* Age 18 or older
* The patient gives written informed consent and can understand the information given
* The patient can participate only once in the study

Exclusion Criteria:

* Earlier resection of the large bowel or rectum
* Active known colitis
* Ileus or gastro-intestinal obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of large bowel cleansing as assessed by the physician performing the colonoscopy. Two validated scoring systems are used.

SECONDARY OUTCOMES:
The subjective grading of patients on ease of taking the large bowel preparation treatment.
Frequency of not completed large bowel preparation treatment.
Frequency of abdominal symptoms due to bowel preparation treatment.
Frequency of incomplete colonoscopies with insufficient view leading to a repeated colonoscopy due to low diagnostic quality at the first attempt.
Costs of large bowel cleansing.
Frequency of abdominal symptoms that start after onset of large bowel preparation treatment and that persists one week after the colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Naredi, MD, PhD, Study Chair — Umeå University; Markku M Haapamaki, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Department of Surgery, Umeå University Hospital, Umeå, Sweden

REFERENCES:
- [Background] Hookey LC, Depew WT, Vanner SJ. Combined low volume polyethylene glycol solution plus stimulant laxatives versus standard volume polyethylene glycol solution: a prospective, randomized study of colon cleansing before colonoscopy. Can J Gastroenterol. 2006 Feb;20(2):101-5. doi: 10.1155/2006/621367. PMID 16482236
- [Result] Haapamaki MM, Lindstrom M, Sandzen B. Low-volume bowel preparation is inferior to standard 4 1 polyethylene glycol. Surg Endosc. 2011 Mar;25(3):897-901. doi: 10.1007/s00464-010-1293-6. Epub 2010 Sep 2. PMID 20812020